CLINICAL TRIAL: NCT02374879
Title: User Performance and System Accuracy Evaluations Using Glucose Adjustment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3128466
Record Dates: First submitted 2015-02-18; First posted 2015-03-02 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Glucose monitoring System (BGMS) (Experimental): Intervention: Blood Glucose monitoring System (BGMS) Results obtained from the BGMS for UP and SA are compared to a reference instrument (YSI)
  Interventions: Device: Blood Glucose Monitoring Systems.

INTERVENTIONS:
Device: Blood Glucose Monitoring Systems. — In vitro diagnostic medical device.

SUMMARY:
This is an open-label, non-randomised pilot study, to evaluate user performance and system accuracy in blood Glucose monitoring system with glucose adjustment. Twelve male and female volunteers aged 18-45, with a documented diagnosis of Type I diabetes for at least 12 will be enrolled in this study.

ELIGIBILITY:
Summary of inclusion criteria.

* Male and female volunteers aged 18-45, with a documented diagnosis of Type I diabetes for at least 12 months and treated with a basal bolus insulin regime, and deemed otherwise healthy as determined by medical history, physical examination, laboratory test values, vital signs and 12-lead ECGs at screening.
* Non-smokers from at least 12 months before study start and for the duration of the study.
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Able to voluntarily provide written informed consent to participate in the study.
* Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol, as confirmed during the informed consent process.
* Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
* The volunteer's primary care physician has confirmed within the last 12 months that there is nothing in their medical history that would preclude their enrolment into a clinical study.
* User Performance Accuracy Testing Only: Self-Monitoring - Volunteer is currently performing unassisted self-monitoring of blood glucose.

Summary of exclusion criteria.

* A severe hypoglycaemic reaction, defined as causing loss of consciousness and/or requiring outside assistance with oral or intravenous glucose or a glucagon injection, within 7 days of the study start date.
* Female volunteers who are pregnant or lactating.
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Current or history of drug or alcohol abuse or a positive drugs of abuse or alcohol test at screening or check-in.
* Participation in a clinical drug study during the 90 days prior to study start.
* Any clinically significant illness within 30 days prior to study start.
* Donation of blood or blood products within 30 days prior to study start, or at any time during the study, except as required by this protocol.
* Weekly alcohol intake exceeding the equivalent of 14 units per week for females or 21 units per week for males.
* Consumption of alcoholic beverages within 48 hours prior to check-in.
* Volunteers with a substantial change in eating habits within 30 days prior to study start or volunteers who cannot comply with the standardised meals proposed for use in the study.
* Prior experience with the BGMSs used for the study.
* Volunteers who are currently working for, have previously worked for, or have an immediate family member working for a company that manufactures or markets blood glucose monitoring products.
* Volunteers who have laboratory training or experience (medical technologist, laboratory technician, laboratory assistant etc).
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
User Performance (UP) evaluation. | Up to 6 hours
  UP evaluation of blood glucose monitoring systems compared to a reference instrument. Samples collected by subject and HCP
System Accuracy (SA) evaluation | Up to 6 hours
  UP evaluation of blood glucose monitoring systems compared to a reference instrument. Samples collected by HCP only.

CONTACTS AND LOCATIONS:
Overall Officials: David J Bell, Principal Investigator — BioKinetic Europe Ltd
Locations (1):
- BioKinetic Europe Ltd, Belfast, Antrim, United Kingdom